CLINICAL TRIAL: NCT00597623
Title: Randomized Double Blind Placebo-controlled Trial of the Efficacy of an Anti-TNF Alpha Agent (Adalimumab, Humira®) in Patients With Incapacitating Hand Osteoarthritis Refractory to Usual Treatment
Brief Title: Efficacy Study of an Anti-Tumor Necrosis Factor (TNF) Alpha Agent in Patients With Hand Osteoarthritis
Acronym: DORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P 051007
Record Dates: First submitted 2008-01-15; First posted 2008-01-18 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-05

CONDITIONS: Hand Osteoarthritis
Keywords: Osteoarthritis; Hand; Tumor Necrosis Factor-alpha inhibitors; Biological Therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 2 injections of Adalimumab (Humira®)
  Interventions: Other: Adalimumab (Humira®)
- 2 (Placebo Comparator): 2 injection of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Adalimumab (Humira®) — syringes for injections under cutaneous dose = 40mg vol = 0.8 ml
  Arms: 1
Other: Placebo — syringes under cutaneous vol = 8 ml
  Arms: 2

SUMMARY:
Digital osteoarthritis (DO) which affects the interphalangeal joints and the Metacarpophalangeal (MCP) of the thumb is a common disease, the prevalence of which increases with age (36% of the population aged over 70). Certain forms of DO with clinical manifestations involving inflammatory features are particularly refractory to usual treatments (analgesics, NSAIDs, braces and local injections). The mechanism of osteoarthritis involves two major cytokines: interleukin-1 beta and tumor necrosis factor alpha. TNF alpha is particularly involved in the inflammation process.

The aim of the present study is to study the efficacy of TNF alpha blockers (2 injections of adalimumab compared to placebo injections in patients with severe and refractory hand osteoarthritis.

We hope that such new therapeutic option may induce substantial pain relief.

DETAILED DESCRIPTION:
Objective: To demonstrate the efficacy of two subcutaneous injections of anti-TNF alpha (adalimumab) in patients with DO refractory to usual treatments (NSAIDs - analgesics).

Design: Randomized placebo-controlled multicenter (20 sites (amendment 18/12/2008)) trial

Trial duration: 6 months follow-up per patient, total trial duration: 12 months

Number of patients: 84(up)

Dose of administration: Two subcutaneous injections separated by a 2-week interval of either adalimumab or placebo. Therapeutic precautions inherent to the prescription of anti-TNF alpha are based upon those recommended in rheumatoid arthritis. With only two injections of anti-TNF alpha, the risk of complications (infectious in particular) inherent to the anti-TNF alpha appears to be extremely slight.

Patient selection: Patients with digital osteoarthritis (DIP and PIP) according to American College of Rheumatology (ACR) criteria (with a recent X-ray, less than 6 months, of the hands, showing signs of digital osteoarthritis), symptomatic for more than 3 months (at least three finger joints) and scored more than 40 mm on a pain visual analog scale (VAS) despite use of a level 1 analgesic (acetaminophen: 4 g daily) andNSAIDs. Main Exclusion criteria are contraindications to anti-TNF alpha according to international guidelines.

Methods: Patients will be seen at a screening visit, then during treatment administration (W0 and W2) and at follow-up visits: W6, 10, 14 and 26. NSAIDs will be stopped at the time of screening.

Efficacy evaluation: The efficacy endpoint is improvement in pain on a pain VAS at different times of assessment (primary endpoint at W6). A more than 50% improvement, in comparison with baseline, will be considered to be significant. Secondary endpoints are: number of tender joints, number of swollen joints, morning stiffness, global assessment of handicap by patient, global assessment of handicap by physician, the DREISER'S algofunctional index, Cochin hand index, weekly evolution of pain ( patient record), and recording of analgesic use (acetaminophen or NSAIDs).

Statistical data: Statistical analysis will be performed on the inter-group difference in the intention-to-treat population. khi-2 will be used only for criteria number 1.

Anticipated result: Significant superiority of adalimumab over placebo which would provide a therapeutic solution in difficult-to-treat patients with hand OA.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-80
* Men or women
* Digital osteoarthritis (DIP and PIP) according to ACR criteria (with recent X-ray, dating from less than 6 months, of the hands showing radiological signs of digital osteoarthritis)
* Symptomatic digital osteoarthritis for more than 3 months (at least every other day) despite taking analgesics and NSAIDs (except when there are contraindications to the latter therapeutic group)
* Osteoarthritis affecting more than three finger joints
* Pain more than 40 mm as evaluated by pain VAS (0-100 mm)
* No contraindication to anti-TNF alpha treatments
* No digital osteoarthritis surgery scheduled within the next 2 months
* Written informed consent

Exclusion Criteria:

* Pregnant women or women of reproductive potential without effective contraception
* Known hypersensitivity
* Patients having already been treated with an anti-TNF alpha
* Finger osteoarthritis secondary to inflammatory rheumatism
* Psoriasis
* Existence of painful syndrome of upper limbs likely to interfere with the monitoring of pain (cervicobrachial neuralgia, incapacitating carpal tunnel syndrome, joint disorders of the elbow or shoulder)
* Inflammatory rheumatism
* Contraindications to anti-TNF alpha agents: patients with suspected reactivation of tuberculosis (phlyctenular IDR, past history of tuberculosis, chest X-ray deemed suspect) or known leukopenia (< 3500 leukocytes), known hepatic cytolysis (transaminases more than twice normal), a history of serious allergy, concomitant infection, past history of serious systemic infection (septicemia), a history of known cancer within the past 5 years, history of multiple sclerosis
* Skin disease incompatible with subcutaneous injection
* Anticoagulant (oral) or treatment with heparin at a curative dose
* Surgery scheduled within the coming 2 months
* Finger surgery scheduled within the coming 6 months
* Local injection of a corticosteroid in a symptomatic finger joint during the previous month
* Local injection of hyaluronic acid in a symptomatic finger joint during the prior 3 months
* Treatment with a slow-acting anti-osteoarthritis agent initiated and colchicine (amendment 26/06/2008) within the previous 3 months
* Oral corticosteroids
* Psychiatric illness
* Non-controlled diabetes "mellitus"
* Known viral hepatitis B or C, HIV infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Level of Pain on visual analogue scale | 4 weeks following the last injection

SECONDARY OUTCOMES:
Number of tender joints | at weeks 4, 6, 10, 14, 26
Number of swollen joints | at weeks 4, 6, 10, 14, 26
Global assessment of handicap by patient | at weeks 4, 6, 10, 14, 26
Global assessment of handicap by physician | at weeks 4, 6, 10, 14, 26
Duration of morning stiffness | at weeks 4, 6, 10, 14, 26
DREISER'S algofunctional index | at weeks 4, 6, 10, 14, 26
Cochin hand index | at weeks 4, 6, 10, 14, 26
Weekly pain recording, and recording of analgesic use (acetaminophen) | at weeks 4, 6, 10, 14, 26
Percentage of non responders according to the number of patients requiring NSAIDS intake during the trial and/or rule out for lack of efficacy | from week 0 until week 26

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Chevalier, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Chevalier X, Ravaud P, Maheu E, Baron G, Rialland A, Vergnaud P, Roux C, Maugars Y, Mulleman D, Lukas C, Wendling D, Lafforgue P, Loeuille D, Foltz V, Richette P; French section of osteoarthritis. Adalimumab in patients with hand osteoarthritis refractory to analgesics and NSAIDs: a randomised, multicentre, double-blind, placebo-controlled trial. Ann Rheum Dis. 2015 Sep;74(9):1697-705. doi: 10.1136/annrheumdis-2014-205348. Epub 2014 May 9. PMID 24817417